CLINICAL TRIAL: NCT03050242
Title: Benefits of Intramuscular Glycopyrrolate Premedication on Intubation With Rigid-videostylet (OptiScope® PM 201, KoMAC Co., Ltd, Seoul, Republic of Korea)
Brief Title: Benefits of Glycopyrrolate on Intubation With Rigid-videostylet (OptiScope®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Clinical Fellow, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017-01-001
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycopyrrolate (Experimental): Glycopyrrolate 0.005mg/kg is administered intramuscularly, one hour before the surgery.
  Interventions: Drug: Glycopyrrolate
- Control (No Intervention): No injection is conducted in this group.

INTERVENTIONS:
Drug: Glycopyrrolate — Intramuscular administration of glycopyrrolate 0.005mg/kg 1 hour before the surgery
  Other Names: intramuscular glycopyrrolate premedication
  Arms: Glycopyrrolate

SUMMARY:
This study is intended to evaluate the efficacy and safety of glycopyrrolate as an antisialagogue prior to intubation with the rigid-videostylet(Optiscope®) in the general anesthesia settings. Upper airway secretions limit the use of the videostylet during during endotracheal intubation. Therefore, in this study, patients will be allocated to either of the two groups according to the administration of glycopyrrolate and the effect of glycopyrrolate in reducing oral secretions will be assessed by the observer while intubating with the rigid-videostylet. The efficacy of the antisialagogic effect on the view during endotracheal intubation will be evaluated.

DETAILED DESCRIPTION:
Recently, the newer forms of intubating devices combining video technologies were introduced. The fiberoptic stylets are useful instrumentations especially for difficult airways and limited neck mobilizations.The OptiScope® is a semi-rigid videostylet designed for endotracheal intubation. While using the device, visualization of the airway might be obscured by the secretions during its insertion. The deterioration of the view leads to intubation failure, resulting in multiple intubation attempts, longer intubating time and desaturation.Therefore, while using the Opticoscope®, proper antisialagogic preparation will be helpful.

Total 78 patients scheduled for general anesthesia aged 20-65 years and Anesthesiologists physical status (ASA) class 1 or 2 will be included. The obese patients (BMI>30) and expected difficult intubation will be excluded. The sample size was estimated based on the preliminary study. With a type Ⅰ error estimate(α) of 0.05 at 80% power, we estimated that 30 patients in each group, or 60 in total, were needed. Considering the drop-out rate of 30%, the total sample size were 78 in total. The patients will be randomly allocated to the glycopyrrolate group(G) and the control group(C). The group-G will received intramuscular glycopyrrolate 0.005mg/kg injection 1 hour before the surgery. For the group-C glycopyrrolate will not be administered. Intubation will be conducted with the OptiScope®. While intubating, the degree of the secretion will be evaluated through the OptiScope® and graded excellent, good, poor and unacceptable according to the dryness and the visualization of the vocal cord. When the vocal cord was seen without secretions, it was stated 'Excellent'. 'Good' was graded when secretions existed without the need for suctioning to visualize the vocal cord. When there were secretions and needed suctioning to clear the view, the subjects were rated 'Poor'. When intubation was failed due to poor visualization of the vocal cord despite the suctioning of the secretion, it was graded 'Unacceptable'. If the intubation is not available within 1 minute, the intubation will be done with the laryngoscope. The time to intubate will be checked by the assist anesthesiologist. The definition of the 'intubation time' is the time between the introduction of the OptiScope® into the mouth and the confirmation of the proper intubation with capnographic wave.The baseline vital signs including systolic blood pressure, mean arterial pressure, diastolic blood pressure and heart rate will be measured before the intubation and 1,3 and 5 minutes after the intubation.

The collected data will be compared with the independent t-test or Mann-Whitney-Wilcoxon test for the continuous variables. Χ2 test and Fisher's exact test will be performed for the categorical variables. Significant level will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic cholecystectomy under general anesthesia
* aged from 19 to 65, adult patients
* american society of anesthesiologist physical status 1,2
* obtaining written informed consent

Exclusion Criteria:

* obese patients with body mass index above 30
* expected difficult intubation (ex. intraoral mass, history of former difficult intubation, limitation of mouth opening..)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
The degree of the secretion | After an average of 1 second from the start of intubation with the OptiScope®.
  The degree of the secretion evaluation done through the OptiScope(R). It was graded by 4-point-scale. Excellent (1) : Dry. No secretion Good (2): Moist Acceptable (2): Wet. Suctioning is NOT required to intubate. Poor(4): Wet. Suctioning is required to intubate

SECONDARY OUTCOMES:
Time to Intubate | 2 minutes after the start of intubation with the OptiScope®.
  It is defined by the time between the introduction of the OptiScope® into the mouth and the confirmation of the proper intubation with capnographic wave.

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho EA, Hwang SH, Lee SH, Ryu KH, Kim YH. Does glycopyrrolate premedication facilitate tracheal intubation with a rigid video-stylet?: A randomized controlled trial. Medicine (Baltimore). 2018 Aug;97(32):e11834. doi: 10.1097/MD.0000000000011834. PMID 30095660